CLINICAL TRIAL: NCT05824975
Title: An Open-label, Multicenter, Dose Escalation and Expansion Phase 1/2 Study to Evaluate the Safety, Tolerability and Pharmacokinetics, and Anti-tumor Activity of GI-102, a CD80-IgG4 Fc-IL-2v Bispecific Fusion Protein, As a Single Agent and in Combination with Conventional Anti-cancer Drugs, Pembrolizumab or Trastuzumab Deruxtecan(T-DXd) in Patients with Advanced or Metastatic Solid Tumors (KEYNOTE-G08)
Brief Title: A Study to Evaluate the Safety and Therapeutic Activity of GI-102 As a Single Agent and in Combination with Conventional Anti-cancer Drugs, Pembrolizumab or Trastuzumab Deruxtecan(T-DXd) in Patients with Advanced Solid Tumors (KEYNOTE-G08)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GI Innovation, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GII-102-P101; KEYNOTE-G08, MK3475-G08 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Soft Tissue Sarcoma (STS); Platinum-resistant Ovarian Cancer (PROC); Hepatocellular Carcinoma (HCC); Colorectal Cancer (CRC); HER2 Negative Breast Cancer; Cutaneous Melanoma; Renal Cell Carcinoma (RCC)
Keywords: GI-102; CD80-IgG4 Fc-IL2 variant; Immunotherapy; IL-2; Interleukin-2; bispecific protein; immunocytokine; CD80; CTLA-4; Pembrolizumab; T-DXd; Trastuzumab deruxtecan; Doxorubicin; Paclitaxel; Bevacizumab; Eribulin
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Carcinoma, Hepatocellular; Colorectal Neoplasms; Melanoma; Carcinoma, Renal Cell; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Doxorubicin; Paclitaxel; Bevacizumab; eribulin; trastuzumab deruxtecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- GI-102 (Experimental): Dose escalation: GI-102 intravenous (IV), multiple ascending doses Dose optimization: GI-102 intravenous (IV), sRP2D Dose optimization: GI-102 intravenous (IV), sRP2D-1 (or sRP2D+1)
  Interventions: Drug: GI-102
- GI-102 subcutaneous (SC) (Experimental): Dose escalation: GI-102 subcutaneous (SC), multiple ascending doses Dose expansion: GI-102 subcutaneous (SC), sRP2D
  Interventions: Drug: GI-102 subcutaneous (SC)
- GI-102 + doxorubicin (Experimental)
  Interventions: Drug: doxorubicin; Drug: GI-102
- GI-102 + paclitaxel + bevacizumab (Experimental)
  Interventions: Drug: paclitaxel; Drug: bevacizumab; Drug: GI-102
- GI-102 + eribulin (Experimental)
  Interventions: Drug: eribulin; Drug: GI-102
- GI-102 + trastuzumab deruxtecan (T-DXd) (Experimental)
  Interventions: Drug: trastuzumab deruxtecan (T-DXd); Drug: GI-102
- GI-102 + pembrolizumab (Experimental)
  Interventions: Drug: pembrolizumab; Drug: GI-102

INTERVENTIONS:
Drug: GI-102 subcutaneous (SC) — 0.12 mg/kg, 0.24 mg/kg or Recommended phase 2 dose of GI-102 will be administered via SC injection Q3W up to 2 years (approximately 35 years).
  Arms: GI-102 subcutaneous (SC)
Drug: GI-102 — Dose level will be escalated from 0.06 mg/kg to 0.45 mg/kg and Recommended phase 2 dose (or RP2D-1, RP2D+1) of GI-102 will be administered via IV infusion Q3W up to 2 years (approximately 35 years).
  Arms: GI-102
Drug: doxorubicin — Doxorubicin will be administered intravenously at a dose of 75 mg/m2 on Day 3 every 3-week (21-day) cycle for up to 6 cycles.
  Arms: GI-102 + doxorubicin
Drug: paclitaxel — Paclitaxel will be administered intravenously over 1 hour at a dose of 80 mg/m2 each time weekly as a diluted solution according to the prescribing information.
  Arms: GI-102 + paclitaxel + bevacizumab
Drug: bevacizumab — Bevacizumab will be administered intravenously at a dose of 10 mg/kg every 2 weeks.
  Arms: GI-102 + paclitaxel + bevacizumab
Drug: eribulin — Eribulin will be administered intravenously at a dose of over 1.4 mg/m2 over 2 to 5 minutes on Days 3 and 10 every 3-week (21-day) cycle.
  Arms: GI-102 + eribulin
Drug: trastuzumab deruxtecan (T-DXd) — T-DXd will be administered initially as a 5.4 mg/kg (or 6.4 mg/kg only for gastric cancer) IV over 30 - 90 minutes every 3 weeks.
  Other Names: ENHERTU®
  Arms: GI-102 + trastuzumab deruxtecan (T-DXd)
Drug: pembrolizumab — pembrolizumab will be administered at a dose of 200 mg as IV infusion Q3W.
  Other Names: KEYTRUDA®
  Arms: GI-102 + pembrolizumab
Drug: GI-102 — Recommended phase 2 dose (or RP2D-1, RP2D-2) of GI-102 will be administered via IV infusion Q3W up to 2 years (approximately 35 years).
  Arms: GI-102 + doxorubicin; GI-102 + eribulin; GI-102 + paclitaxel + bevacizumab; GI-102 + pembrolizumab; GI-102 + trastuzumab deruxtecan (T-DXd)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and therapeutic activity of GI-102 as a single agent and in combination with conventional anti-cancer drugs, pembrolizumab or trastuzumab deruxtecan(T-DXd) over a range of advanced and/or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, and anti-tumor effect of GI-102 as a single agent and in combination with conventional anti-cancer drugs, pembrolizumab or trastuzumab deruxtecan(T-DXd) over a range of advanced and/or metastatic solid tumors. This study is adaptive in nature.

The study is composed of four parts:

* Part A: Dose escalation and optimization phase of GI-102 intravenous (IV) monotherapy

  * Part A dose escalation phase
  * Part A dose optimization phase: Dose optimization cohorts in patients with 2L+, CPI-refractory metastatic melanoma
* Part B: Dose escalation and expansion phase of GI-102 subcutaneous (SC) monotherapy
* Part C: Indication specific cohorts of GI-102 IV in combination with conventional anti-cancer drugs or trastuzumab deruxtecan (T-DXd)
* Part D: Indication specific cohorts of GI-102 IV in combination with pembrolizumab

GI-102 is a novel bi-specific Fc fusion protein containing the CD80 ectodomain as an N-terminal moiety and an interleukin (IL)-2 variant as a C-terminal moiety configurated via a human immunoglobulin G4 (IgG4) Fc. GI-102 has unique characteristics by having bispecificity to CD80 and IL2Rβγ. The CD80 portion is responsible for targeting tumor/immune cells while blocking CTLA-4 expressed on the Treg cells. The IL-2v of GI-102 is designed to abolish IL-2Rα affinity and therefore minimize the effect on Treg while it has very outstanding effect on NK and CD8 T cell proliferation and activity through IL-2Rbr affinity.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females aged ≥ 18 years (or ≥ 19 years according to local regulatory guidelines) at the time of screening.
* Has adequate organ and marrow function as defined in protocol.
* Measurable disease as per RECIST v1.1.
* ECOG performance status 0-1.
* Adverse events related to any prior chemotherapy, radiotherapy, immunotherapy, other prior systemic anti-cancer therapy, or surgery must have resolved to Grade ≤1, except alopecia and Grade 2 peripheral neuropathy.
* HIV infected patients must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease as defined in protocol.

Key Exclusion Criteria:

* Has known active CNS metastases and/or carcinomatous meningitis.
* An active second malignancy.
* Has active or a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has active tuberculosis or has a known history of active tuberculosis.
* Active or uncontrolled infections, or severe infection within 4 weeks before study treatment administration.
* History of chronic liver disease or evidence of hepatic cirrhosis, except patients with liver metastasis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Previous immunotherapies related to mode of action of GI-102.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive medications within 2 weeks prior to Cycle 1 Day 1.
* Administration of prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment.
* Radiotherapy within the last 2 weeks before start of study treatment administration, with exception of limited field palliative radiotherapy.
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1.
* Known hypersensitivity to any of the components of the drug products and/or excipients of GI-102.

Other protocol defined inclusion exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of Dose-Limiting Toxicity (DLTs) (dose escalation phase of Part A and B) | Study Day 1, assessed up to DLT period (3 weeks after treatment)
  A DLT is defined as a clinically significant AE (classified according to the NCI CTCAE version 5) or significant laboratory abnormality that occur during the DLT assessment periods, during dose escalation and dose expansion, and is considered by the Investigator to be related to GI-102.
Incidence, nature, and severity of adverse events (AEs) and immune-related AEs (irAEs) (dose escalation phase of Part A and B) | Study Day 1, assessed up to approximately 24 months
  An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. All AE events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Objective Response Rate (ORR) (dose optimization phase of Part A, dose expansion phase of Part B, Part C and D) | Study Day 1, assessed up to approximately 24 months
  ORR is defined as the percentage of participants with investigator-assessed objective response of complete response (CR) or partial response (PR). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (dose escalation phase of Part A and B) | Study Day 1, assessed up to approximately 24 months
  ORR is defined as the percentage of participants with investigator-assessed objective response of complete response (CR) or partial response (PR). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).
Incidence and nature of Dose-Limiting Toxicity (DLTs) (dose optimization phase of Part A, dose expansion phase of Part B, Part C and D) | Study Day 1, assessed up to DLT period (3 weeks after treatment)
  A DLT is defined as a clinically significant AE (classified according to the NCI CTCAE version 5) or significant laboratory abnormality that occur during the DLT assessment periods, during dose escalation and dose expansion, and is considered by the Investigator to be related to GI-102.
Incidence, nature, and severity of adverse events (AEs) and immune-related AEs (irAEs) (dose optimization phase of Part A, dose expansion phase of Part B, Part C and D) | Study Day 1, assessed up to approximately 24 months
  An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. All AE events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Disease Control Rate (DCR) | Study Day 1, assessed up to approximately 24 months
  DCR is defined as the percentage of patients who have achieved CR, PR and stable disease (SD), per RECIST v1.1 guideline as determined by the investigators.
Duration of objective response (DoR) | Study Day 1, assessed up to approximately 24 months
  DCR is defined as the time from the first occurrence of a documented objective response to the time of the first document disease progression or death from any cause, whichever occurs first, per RECIST v1.1 as determined by the investigator.
Progression-free survival (PFS) | 6-month, 12-month, and 18-month
  PFS is defined as the time from the first study treatment (Day 1) to the first occurrence of progression or death from any cause, whichever occurs first, per RECIST v1.1 guideline as determined by the investigator
Overall survival (OS) | 12-month and 18-month
  OS is defined as the time from the first study treatment to death from any cause
Peak plasma concentration (Cmax) of GI-102 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Half-life of GI-102 (T1/2) | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Area under the plasma concentration versus time curve (AUC) of GI-102 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Clearance of GI-102 | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level
Volume of distribution (Vd) of GI-102 after administration | Study Day 1, assessed up to approximately 24 months
  Based on the concentration vs time profile by dose level

OTHER OUTCOMES:
Incidence of anti-GI-102 antibody (ADA) and neutralizing antibody (Nab) | Study Day 1, assessed up to approximately 24 months
  Serum will be assessed for the presence of ADA and Nab based on the appropriate assay.
Immunophenotyping of peripheral blood CD4+ T cells | Study Day 1, assessed up to approximately 24 months
  CD4+ T cells in peripheral blood will be assessed by flow cytometry at various time points
Immunophenotyping of peripheral blood CD8+ T cells | Study Day 1, assessed up to approximately 24 months
  CD8+ T cells in peripheral blood will be assessed by flow cytometry at various time points
Immunophenotyping of peripheral blood Treg cells | Study Day 1, assessed up to approximately 24 months
  Treg cells in peripheral blood will be assessed by flow cytometry at various time points

CONTACTS AND LOCATIONS:
Overall Officials: Nari Yun, PhD, Study Director — GI Innovation, Inc.
Locations (10):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Minnesota, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- South Korea (5):
  - Seoul National University Hospital, Seoul, Seoul
  - St. Vincent's Hospital, Suwon, suwon
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No